CLINICAL TRIAL: NCT00390247
Title: Thalidomide for the Treatment of Malnutrition Inflammation Syndrome in Peritoneal Dialysis Patients: A Randomized Control Trial
Brief Title: Thalidomide for the Treatment of Malnutrition Inflammation Syndrome in Peritoneal Dialysis Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Fail of applying funding
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRE-2006.291
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2007-04

CONDITIONS: Peritoneal Dialysis; Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Thalidomide

INTERVENTIONS:
Drug: thalidomide

SUMMARY:
Hypothesis In peritoneal dialysis (PD) patients, malnutrition, inflammation and atherosclerotic cardiovascular disease commonly coexist. The triad has been coined the "MIA syndrome". Proinflammatory cytokines, such as tumor necrosis factor-alpha (TNF-alpha), plays a central role in the pathogenesis of the MIA syndrome. Thalidomide selectively inhibits the production of TNF-alpha and represents a valuable anti-cytokine therapy.

Specific Aim To study the effect of thalidomide in attenuating or reversing malnutrition and systemic inflammation in PD patients.

Research Plan

Design: Double-blinded randomised prospective placebo control trial. Setting: Renal unit of a university teaching hospital. Subjects: Sixty prevalent PD patients with evidence of malnutrition. Interventions: Patients will be randomised to receive either oral thalidomide 100 mg nocte or placebo.

Main outcome measures: Patients will be followed for 1 year. Nutritional parameters including serum albumin, subjective global assessment, malnutrition-inflammation score, normalised protein nitrogen appearance, fat-free edema-free body mass and anthropometry measurements will be monitored. Systemic inflammatory markers such as serum C-reactive protein and IL-6 will be assayed. Hospitalisation, cardiovascular events, and overall patient survival will also be compared during study period.

Expected Outcome

Nutritional parameters and markers of systemic inflammation are expected to improve with thalidomide therapy. The magnitude of improvement in nutrition, as well as patient morbidity, will be compared with placebo.

In Hong Kong, 80% of end-stage renal failure patients are treated with PD. Malnutrition, cardiovascular disease and systemic inflammatory response are all common in our clinical practice. They are major causes of patient morbidity and mortality. As a readily available anti-cytokine therapy, thalidomide may represent a valuable treatment of the MIA syndrome. The proposed study will provide important insight on the clinical benefit of thalidomide treatment in malnourished PD patients, which accounts for about one-third of our dialysis population.

DETAILED DESCRIPTION:
Overall study design

This is a single-center randomized placebo control study on 60 prevalent PD patients.

Recruitment phase will take up to 12 months, and the study phase will be 1 year. Study code will only be revealed at the end of the study period or if patients develop serious adverse reactions.

Patient selection

A randomized prospective study will be performed in 60 stable PD patients. Recruitment criteria are:

A. clinically stable adult patients (18 to 80 years old) on PD; and

B. evidence of malnutrition:

1. overall subjective global assessment score < 5; or
2. malnutrition inflammation score > 9; or
3. serum albumin < 35 g/L C. written patient informed consent

   Exclusion criteria are:

   Patients who are planned to have elective living donor transplant within 6 months Patients who are planned to transfer to other renal center within 6 months High likelihood of early withdrawal from the study (e.g. myocardial infarction, severe or unstable coronary disease, stroke, severe liver disease within 3 months) Active infection or systemic inflammatory disease. Current malignant disease Pregnancy or breast-feeding Women of childbearing potential with unreliable birth control methods Known hypersensitivity to thalidomide

   Baseline data including age, sex, underlying renal disease, presence of diabetes, hepatitis B status, requirement of helper for dialysis procedure, PD regimen and duration on dialysis are recorded.

   Interventions

   After initial evaluation in a screening visit at -4 week, patients will be randomly assigned to receive either oral thalidomide 100 mg nocte or placebo. Thalidomide will be obtained from Penn Pharmaceuticals Ltd (Gwent, UK) as 100 mg tablets, and prescribed in accordance with the published guidelines for the clinical use and dispensing of thalidomide [34]. There will be 30 patients on each arm of randomization. Dialysis prescription will be changed only if there is clinical evidence of underdialysis. Both patients and investigators will be blinded from the therapy during follow up assessment. Side effects will be recorded and the drug will be discontinued when clinically necessary.

   Clinical follow up

   Patients will be followed at at -4 (screening), 0, 4, 8, 12, 18, 24, 30, 36, 44 and 52 weeks. The following clinical data will be documented during each visit:

   Body height and body weight Blood pressure Compliance to thalidomide by pill count Compliance to dialysis exchange by direct questioning Skin itchiness score from 0 to 3+, as described previously [31]

   Body-mass index and body surface area will be computed. The majority of patients will be on three or four 2-liter exchanges per day. Blood pressure or edema are controlled with standard anti-hypertensive agents and/or hypertonic dialysate.

   Laboratory parameters

   A full panel of biochemical parameters will be monitored:

   Hemoglobin, plasma sodium, potassium, urea, creatinine, albumin, calcium, phosphate, alkaline phosphatase, and alanine transaminase at -4, 0, 4, 8, 12, 18, 24, 30, 36, 44 and 52 weeks Fasting serum glucose, lipid and iron profile at 0, 24 and 52 weeks Serum parathyroid hormone at 0 and 52 weeks Serum inflammatory markers at 0, 12, 24, 36 and 52 weeks

   Inflammatory markers include serum C-reactive protein (CRP), interleukin-6 (IL-6), leptin, adiponectin, tumor necrosis factor alpha (TNF-alpha) and fibrinogen levels, as suggested by other groups [35-38].

   Nutritional assessment

   Nutritional status will assessed by subjective global assessment (SGA), comprehensive malnutrition-inflammation score (MIS), normalized protein nitrogen appearance (NPNA), serum albumin level, anthropometric lean body mass (LBM), and fat-free edema-free body mass (FEBM).

   SGA will be performed at -4, 0, 12, 24, 36 and 52 weeks by a single observer. The 4-item 7-point scoring system proposed by Enia et al [39] will be used. MIS will be performed at -4, 0, 12, 24, 36 and 52 weeks. The calculation of MIS has been described previously [40]. Briefly, MIS consists of 4 main parts and 10 components, all scored from 0 (normal) to 3 (very severe). The total score ranges from 0 to 30.

   FEBM and PNA will be measured by creatinine kinetics at 0, 24 and 52 weeks. A 24-hour dialysate and urine collections will be performed. Total and peritoneal Kt/V are determined by standard methods. Residual GFR is calculated as average of 24-hour urinary urea and creatinine clearance. FEBM is calculated according to the formula of Forbes and Brunining [41]. PNA is derived from the Randerson's formula [42]. It is further normalized to standard body weight.

   Anthropometric measurements will be performed at 0, 12, 24, 36 and 52 weeks by a single observer. This include bicep, tricep, subscapular and supra-iliac skin fold thickness, and midarm muscle circumference. Derived variables by anthropometric measurements, including lean body mass (LBM) and percentage of body fat, will be computed by standard formula [43].

   Pulse wave velocity

   Pulse wave velocity (PWV), an index of aortic stiffness, is measured using an automatic computerized recorder at 0, 24 and 52 weeks. The results will be analyzed by the Complior SP program (Artech Medical, France). Briefly, pressure-sensitive transducers are placed over the neck (carotid artery), wrist (radial artery) and groin (femoral artery) with the patient in the supine position on day of haemodialysis treatment before putting patient to the dialysis machine. PWV of the carotid-femoral and carotid-radial territory is calculated by dividing the distance between the sensors by the time corresponding to the period separating the start of the rising phase of the carotid pulse wave and that of the femoral and also the radial pulse waves. The procedure takes 10 to15 seconds to complete. The test will be performed by the same observer to eliminate effect of intra-observer variation.

   Health-related quality of life

   Patient acceptance and satisfaction will be assessed by the Chinese translation of "Kidney Disease Quality of Life Short Form (KDQOL-SFTM), version 1.3", at 0 and 52 weeks.

   Outcome

   The major outcome measure is nutritional status, as detailed above. The schedule of various tests is summarized in Appendix 2. Secondary outcomes include the followings:

   Change in arterial pulse wave velocity Total number of days of hospital admission during study period Composite cardiovascular end point: cardiovascular death, non-fatal myocardial infarction or stroke, hospital admission for unstable angina, coronary intervention, transient ischemic attack, or lower limb ischemia Number of episode of peritonitis during study period All cause mortality

   Transplantation, conversion to hemodialysis, recovery of renal function, and transfer out of the unit will also be recorded.
4. Potential Outcomes

In Hong Kong, 80% of end-stage renal failure patients are treated with peritoneal dialysis (PD). In 2004, there were over 3000 PD patients in Hong Kong. Malnutrition, cardiovascular disease and systemic inflammatory state are all common in our clinical practice. They are major causes of patient morbidity and mortality. The financial implication is considerable.

As a readily available anti-cytokine therapy, thalidomide may represent a valuable treatment of the MIA syndrome. The proposed study will provide important insight on the clinical benefit of thalidomide treatment in malnourished PD patients, which accounts for about one-third of our dialysis population.

Data Analysis

Statistical analysis will be performed by SPSS for Windows software version 11.5 (SPSS Inc., Chicago, IL). All data will be expressed in mean +/- standard deviation unless otherwise specified. Serial changes of nutritional parameters, dialysis adequacy, and inflammatory markers will be compared to the baseline values by analysis of variance for multiple measures (MANOVA). Serial change in residual GFR is examined by Wilcoxon's rank sum test with Bonferroni's correction for multiple comparison because of skewed data. Nutritional status and systemic inflammatory markers after one year will be compared between the 2 groups by Student's t-test for parametric data. Hospitalization and peritonitis rate between the groups are compared by Kruskal-Wallis test because the data will be highly skewed. Actuarial patient survival will be compared by logrank test with Kaplan-Meier survival curves and treatment group as stratifying variable.

ELIGIBILITY:
Inclusion Criteria:

A. clinically stable adult patients (18 to 80 years old) on PD; and

B. evidence of malnutrition:

1. overall subjective global assessment score < 5; or
2. malnutrition inflammation score > 9; or
3. serum albumin < 35 g/L C. written patient informed consent

Exclusion Criteria:

Patients who are planned to have elective living donor transplant within 6 months Patients who are planned to transfer to other renal center within 6 months High likelihood of early withdrawal from the study (e.g. myocardial infarction, severe or unstable coronary disease, stroke, severe liver disease within 3 months) Active infection or systemic inflammatory disease. Current malignant disease Pregnancy or breast-feeding Women of childbearing potential with unreliable birth control methods Known hypersensitivity to thalidomide

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | 12 months

SECONDARY OUTCOMES:
Change in arterial pulse wave velocity | 12 months
Total number of days of hospital admission during study period | 12 months
Composite cardiovascular end point | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Cheuk-Chun Szeto, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Renal Unit, Department of Medicine & Therapeutics, Prince of Wales Hospital, Hong Kong, Hong Kong